CLINICAL TRIAL: NCT02150733
Title: A Phase 1, Open-Label Study Assessing the Impact of Hepatic Impairment on the Pharmacokinetics of Tivantinib in Subjects With Advanced Solid Tumors
Brief Title: Pharmacokinetics of Tivantinib in Subjects With Advanced Solid Tumors and Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ197-A-U160
Record Dates: First submitted 2014-05-20; First posted 2014-05-30 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-07

CONDITIONS: Hepatic Impairment; Solid Tumor; Cancer
MeSH Terms: conditions — Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - Normal hepatic function (Experimental): Subjects with normal hepatic function
  Interventions: Drug: Tivantinib
- Group 2 - Mild hepatic impairment (Experimental): Subjects with mild hepatic impairment by Child-Pugh classification scores
  Interventions: Drug: Tivantinib
- Group 3 - Moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment by Child-Pugh classification scores
  Interventions: Drug: Tivantinib
- Group 4 - Severe hepatic impairment (Experimental): Subjects with severe hepatic impairment by Child-Pugh classification scores
  Interventions: Drug: Tivantinib

INTERVENTIONS:
Drug: Tivantinib — Single oral administration of Tivantinib 120 mg on Day 1 followed by Tivantinib 360 mg twice daily in the extension phase.
  Arms: Group 1 - Normal hepatic function
Drug: Tivantinib — Single oral administration of Tivantinib 120 mg on Day 1 followed by Tivantinib 120 mg twice daily in the extension phase
  Arms: Group 2 - Mild hepatic impairment
Drug: Tivantinib — Single oral administration of Tivantinib 120 mg on Day 1 followed by Tivantinib 120 mg once daily in the extension phase
  Arms: Group 3 - Moderate hepatic impairment
Drug: Tivantinib — Single oral administration of Tivantinib 120 mg on Day 1 followed by Tivantinib 120 mg once every other day in the extension phase
  Arms: Group 4 - Severe hepatic impairment

SUMMARY:
This is a multi-center, open-label, Phase 1 study to evaluate the impact of hepatic impairment on the pharmacokinetics of Tivantinib in cancer subjects with varying degrees of hepatic function, from normal to severely impaired.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed advanced solid tumor. However, Hepatocellular Carcinoma (HCC) subjects are allowed without histological confirmation as long as there is radiological diagnosis as per standard criteria
2. Male or female ≥18 years of age
3. Life expectancy of >12 weeks
4. Women of childbearing potential (WOCBP) must have a negative pregnancy test performed prior to the start of study drug
5. Male subjects and WOCBP must agree to use double barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug
6. Subjects with impaired hepatic function will be grouped according to Child-Pugh classification score
7. Subjects with biliary obstruction for whom a biliary drain or stent has been placed are eligible, provided that the drain or stent has been in place for at least 10 days prior to the first dose of Tivantinib, and the subject's liver function has stabilized as defined by 2 measurements at least 5 days apart that put the subject in the same hepatic impairment group
8. Eastern Cooperative Oncology Group (ECOG) performance status ≥2
9. Adequate bone marrow and renal function
10. Ability to provide written informed consent, comply with protocol visits and procedures, take oral medication, and not have any active infection or chronic comorbidity that would interfere with therapy
11. Fully informed about their illness and the investigational nature of the study protocol and must sign and date an Institutional Review Board-approved Informed Consent Form

Exclusion Criteria:

1. History of liver transplant
2. Any major surgical procedure within 3 weeks prior to the first dose of study drug;
3. Active, clinically serious infections defined as ≥Grade 2 according to NCI Common Toxicity Criteria for Adverse Effects (CTCAE), version 4.0
4. Known metastatic brain or meningeal tumors, unless the subject is >3 months from definitive therapy and clinically stable (supportive therapy with steroids or anticonvulsant medications is allowed) with respect to the tumor at the time of the first dose of study drug
5. History of cardiac disease

   * Active coronary artery disease, defined as myocardial infarction, unstable angina, coronary bypass graft, or stenting within 6 months prior to study entry
   * Evidence of uncontrolled bradycardia or other cardiac arrhythmia defined as ≥Grade 2 according to NCI CTCAE, version 4.0, or uncontrolled hypertension
6. Any condition that is unstable or that could jeopardize the safety of the subject and the subject's protocol compliance, including known infection with human immunodeficiency virus
7. Significant gastrointestinal disorders, in the opinion of the Investigator
8. Pregnant or breastfeeding
9. Received Tivantinib as prior therapy
10. Received anti-cancer therapy, including antibody, retinoid, or hormonal treatment (except megestrol acetate as supportive care), and radiation, within 3 weeks before dosing. Prior and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin and analogs for neuroendocrine tumors are permitted
11. Any other investigational drug/medical device within 3 weeks prior to the first dose
12. Substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results
13. Subjects receiving Coumadin anticoagulants
14. Inability to swallow oral medications
15. Administration or possibility of initiating or continuing any treatment with any known Cytochrome P450 3A4 (CYP3A4) and CYP2C19 enzyme and P-glycoprotein altering drugs (inducer or inhibitor) or non drug agents within 14 days prior to dosing and during the primary objective phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetic parameters of Tivantinib | 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours after a single dose and 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after Cycle 1 Day 11 dose
  The following pharmacokinetic parameters will be determined: population estimates of apparent total clearance (CL/F), apparent volume of distribution (V/F), area under the concentration-time curve during the dosing interval (AUCtau), and maximum concentration (Cmax) during the dosing interval.

SECONDARY OUTCOMES:
Composite of plasma pharmacokinetic parameters of Tivantinib | 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours after a single dose and 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after Cycle 1 Day 11 dose
  The following pharmacokinetic parameters will be determined: area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) and Cmax after single dose, time to maximum plasma concentration (Tmax)
Composite of plasma pharmacokinetic parameters of Tivantinib metabolites | 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours after a single dose and 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after Cycle 1 Day 11 dose]
  The following pharmacokinetic parameters will be determined: Cmax and AUClast, AUCtau, Tmax, and metabolite ratios for Cmax, AUClast, and AUCtau.

CONTACTS AND LOCATIONS:
Overall Officials: Masaya Tachibana, PhD, Study Director — Daiichi Sankyo
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/